CLINICAL TRIAL: NCT07155408
Title: The Effect of Combined Use of Povidone-Iodine and Rifampicin on Wound Healing and Infection Prevention in Scalp Antisepsis for Hair Transplantation
Brief Title: Combined Use of Povidone-Iodine and Rifampicin in Hair Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elif Asena KANTARCI (Other)
Responsible Party: Sponsor-Investigator, Elif Asena KANTARCI, Lecturer, Vocational School of Health Services, Bahçeşehir University
Organization: Bahçeşehir University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAU-EAS-2025-001; E-22481095-020-1516 (Other: Bahcesehir University Clinical Research Ethics Committee)
Record Dates: First submitted 2025-08-14; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Androgenetic Alopecia; Wound Healing
Keywords: Androgenetic Alopecia; Povidone-Iodine; Rifampicin; Wound Healing; Scalp Antisepsis; Postoperative Care; Hair Transplantation
MeSH Terms: conditions — Alopecia | interventions — Povidone-Iodine; Rifampin

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to two parallel groups: one receiving the standard povidone-iodine antisepsis protocol and the other receiving the combined povidone-iodine and rifampicin protocol. Outcomes were measured simultaneously in both groups.
Masking Description: Due to the visible nature of antiseptic application methods, no blinding was performed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Povidone-Iodine Antisepsis Protocol (Active Comparator): Participants receive preoperative skin antisepsis using the standard povidone-iodine protocol. The antiseptic is applied according to standard surgical preparation guidelines prior to hair transplantation procedures. Outcomes are measured postoperatively following the standard clinical follow-up schedule.
  Interventions: Drug: Povidone-Iodine 10%
- Combined Povidone-Iodine and Rifampicin Protocol (Experimental): Participants receive preoperative skin antisepsis using a combination of povidone-iodine and rifampicin solution. The antiseptic mixture is applied according to study-specific preparation guidelines prior to hair transplantation procedures. Outcomes are measured postoperatively following the standard clinical follow-up schedule.
  Interventions: Drug: Povidone-Iodine 10%; Drug: Povidone-Iodine + Rifampicin

INTERVENTIONS:
Drug: Povidone-Iodine 10% — Preoperative skin antisepsis performed with 10% povidone-iodine solution according to standard surgical preparation guidelines before hair transplantation.
Drug: Povidone-Iodine + Rifampicin — Preoperative skin antisepsis performed with a combination of 10% povidone-iodine and rifampicin solution according to study-specific preparation guidelines before hair transplantation.
  Arms: Combined Povidone-Iodine and Rifampicin Protocol

SUMMARY:
This randomized controlled clinical trial was designed to evaluate the effectiveness of combining 10% povidone-iodine with 125 mg rifampicin for preoperative scalp antisepsis in hair transplantation procedures. The study was conducted in a private hair transplantation clinic between December 2021 and May 2022. A total of 65 adult patients meeting the inclusion criteria were enrolled and randomly assigned to one of two groups: the experimental group (n=34), which received the combined povidone-iodine plus rifampicin protocol, and the control group (n=31), which received povidone-iodine alone as the standard preoperative antisepsis protocol.

Data collection included the use of standardized forms, intraoperative and postoperative observation records, and photographic documentation. Follow-up assessments were performed on postoperative days 3, 7, and 14. The primary aim of the study was to assess the potential of this combined antiseptic protocol to improve wound care and infection prevention practices in hair transplantation surgery.

DETAILED DESCRIPTION:
This study was designed to evaluate the effect of the combined use of povidone-iodine and rifampicin for scalp antisepsis in hair transplantation. The study employed a randomized controlled design, involving adult patients undergoing elective hair transplantation procedures. Participants were randomly assigned to an experimental group receiving the combined antisepsis protocol or a control group receiving standard povidone-iodine alone.

The inclusion criteria included patients over 18 years of age, undergoing elective hair transplantation, and providing informed consent. Exclusion criteria included hypersensitivity to the antiseptic agents or active dermatological conditions on the scalp.

The antiseptic agents were applied preoperatively before the transplantation procedure. Patients were monitored postoperatively at scheduled intervals, and the antisepsis process was documented using standardized photographic assessments.

The total sample included 65 patients. The study duration involved approximately 14 days of follow-up. No interim analysis was conducted. The study protocol was approved by the Bahcesehir University Clinical Research Ethics Committee.

This clinical protocol aims to contribute to the evidence base regarding the use of combination antiseptic protocols in minor surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Individuals scheduled for hair transplantation surgery
* Fitzpatrick skin type between I and IV
* Willingness to participate and sign the written informed consent form
* Overall health status suitable for the procedure (after preoperative evaluation)

Exclusion Criteria:

* Presence of active infection, open wound, or dermatological disease at the surgical site
* Systemic infection or immunosuppressive disorders
* Known allergy or sensitivity to povidone-iodine or rifampicin
* Bleeding disorders or current use of anticoagulant therapy
* Pregnancy or breastfeeding
* History of hair transplantation or similar surgical procedure within the last 6 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Postoperative wound infection rate | Within 14 days post-operation
  Incidence of clinically diagnosed postoperative wound infection, defined by the presence of redness, swelling, tenderness, purulent discharge, or positive bacterial culture, following hair transplantation procedures. Infection will be confirmed based on clinical examination by a qualified physician.

SECONDARY OUTCOMES:
Wound healing time | Assessed daily until complete epithelialization, up to 14 days post-operation.
  Number of days required for complete epithelialization of the donor and recipient sites, assessed by visual inspection and patient report. Complete epithelialization is defined as the absence of open wound areas and formation of intact skin.
Postoperative pain score | 24 hours, 72 hours, and 7 days post-operation.
  Pain intensity reported by the patient using a Visual Analog Scale (VAS) from 0 (no pain) to 10 (worst possible pain) at donor and recipient sites.
Postoperative erythema score | 24 hours, 72 hours, and 7 days post-operation.
  Degree of redness at the donor and recipient sites, scored by the investigator using a standardized erythema grading scale (0-3, where 0 = none, 3 = severe).
Incidence of allergic or hypersensitivity reactions | Within 14 days post-operation.
  Number of patients developing localized or systemic hypersensitivity reactions (e.g., rash, itching, swelling, anaphylaxis) following application of antiseptic solutions.

CONTACTS AND LOCATIONS:
Overall Officials: Fadime ÇINAR, Assoc. Prof.,PhD, Study Chair — Nisantasi University, School of Health Sciences, Department of Nursing
Locations (1):
- Bahcesehir University, School of Health Sciences, Department of Nursing, Istanbul, Besiktas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared for this study. Due to privacy considerations, institutional policies, and ethical regulations, a data sharing plan has not been developed.